CLINICAL TRIAL: NCT00330278
Title: A Randomized, Double-Blind, Placebo Controlled Trial of Cefazolin Given Either 30 Minutes Prior to Cesarean Section or at Cord Clamping
Brief Title: Timing of Prophylactic Antibiotics for Cesarean Sections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HR # 11120
Record Dates: First submitted 2006-05-25; First posted 2006-05-26 (Estimated); Last update posted 2007-09-27 (Estimated); Status verified 2006-01

CONDITIONS: Endometritis; Wound Infection
Keywords: Cesarean section; Antibiotic prophylaxis; Cefazolin
MeSH Terms: conditions — Endometritis; Wound Infection | interventions — Cefazolin

INTERVENTIONS:
Drug: Cefazolin

SUMMARY:
This is a randomized, double-blinded placebo controlled trial of cefazolin timing before cesarean section fo infection prophylaxis. Subjects are randomized to cefazolin either 30 minutes prior to skin incision or at time of cord-clamping. Primary outcome is infectious morbidity including wound infections and endometritis.

ELIGIBILITY:
Inclusion Criteria:

Pregnant 24-43 weeks gestation > 18 years old Requiring cesarean section -

Exclusion Criteria:

Receiving antibiotics < 18 years old Allergy to cefazolin

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 350
Dates: Start 2003-01; Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Combined infectious morbidity - endometritis + wound infection

SECONDARY OUTCOMES:
Neonatal sepsis
Allergic reactions

CONTACTS AND LOCATIONS:
Overall Officials: Scott A Sullivan, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States